CLINICAL TRIAL: NCT02884258
Title: In Vitro Fertilization (IVF) Outcome After Bariatric Surgery: a Multicentric Case-control Study.
Brief Title: IVF Outcome After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Clinique Mathilde (Other)
Responsible Party: Sponsor
Other Study IDs: IVF after Bariatric surgery
Record Dates: First submitted 2016-07-26; First posted 2016-08-30 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Infertility; Obesity
Keywords: Assisted Reproductive Technology; Obesity; Bariatric Surgery; Infertility; Fertility Preservation
MeSH Terms: conditions — Infertility; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Bariatric surgery group: Women undergoing IVF (IVF or ICSI) with a history of bariatric surgery (surgery procedures include sleeve gastrectomies and by-passes). No intervention is involved.
- Control Group: 1. Women undergoing IVF with no history of bariatric surgery and matched to bariatric surgery patients for weight, parity and age. 2. non-operated severely obese women

SUMMARY:
This case-control study compares IVF results and live birth rates in women undergoing IVF with a history of bariatric surgery as compared to 2 age-matched control groups composed of (A) non-operated women matched on cases' post-operative BMI (controls 1) and (B) non-operated severely obese women (controls 2).

DETAILED DESCRIPTION:
A preliminary study in the participating center showed a trend to lower ovarian response to stimulation and live birth rates after bariatric surgery compared to weight-matched patients. However, statistical significance was not reached, as the sample size was small.

The aim of the research project is to study the ovarian response and live birth rates of this bariatric surgery population, with a sufficient number of patients, in order to reach higher statistical power. This case-control study will involve 3 IVF (in-vitro fertilization) centers in France . All patients undergoing IVF with a history of bariatric surgery will be included from January 2012. Each case will be matched for BMI and age to the 2 next patients without bariatric surgery history and undergoing IVF and to one non-operated severely obese woman. Surgery procedures include sleeve gastrectomies and by-passes. The IVF results and live birth rates will be compared between the three groups.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing IVF and with a history of bariatric surgery

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women underoing IVF and having undergone bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2012-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Live birth rates | nine months after embryo transfer
  number of live births divided by the number of embryo transfers

SECONDARY OUTCOMES:
average number of mature oocytes obtained | The day of oocyte retrieval in the case of IVF with sperm injection (ICSI) just after decoronisation, or on day one after oocyte retrieval in classical IVF. Oocyte retrieval occurs 36 hours after hCG injection after an ovarian stimulation protocol.
  the average number of mature oocytes obtained per IVF cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Mathilde, Rouen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grzegorczyk-Martin V, Freour T, De Bantel Finet A, Bonnet E, Merzouk M, Roset J, Roger V, Cedrin-Durnerin I, Wainer R, Avril C, Landais P. IVF outcomes in patients with a history of bariatric surgery: a multicenter retrospective cohort study. Hum Reprod. 2020 Dec 1;35(12):2755-2762. doi: 10.1093/humrep/deaa208. PMID 33083823